CLINICAL TRIAL: NCT05108116
Title: Phenotyping the Alignment and Rotational Parameters of the Lower Limb in Young Non-osteoarthritic Population
Brief Title: Phenotyping the Alignment of the Lower Limb
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: UP-CC-Ortho-LLimbAlign
Record Dates: First submitted 2021-10-12; First posted 2021-11-04 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Lower Limb Deformity
Keywords: EOS 2D/3D; Lower limb alignment; Lower limb rotation; Osteoarthritis of the Knee; Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 18-30 year-old, healthy volunteers
  * Age: 18-30 years
  * BMI: <30
  * No previous surgery on lower limb or spine
  * No known developmental disorder
  * Without any orthopaedic complaint
  Interventions: Diagnostic Test: EOS

INTERVENTIONS:
Diagnostic Test: EOS — EOS Micro Dose imaging will be done. SterEOS 3D recontruction of the lower limb and pelvis will be performed.
  Other Names: EOS 2D/3D scanning and SterEOS 3D reconstruction

SUMMARY:
In the international literature there are only few publication about the normal biomechanical parameters of the lower limb examined prospectively in healthy population. The goal of our study to determine 15 anatomical and biomechanical parameters of the lower limb using 3D reconstruction based on upright, stereo radiographs in young, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 years
* BMI: < 30
* Without orthopaedic complaint

Exclusion Criteria:

* Previous surgery on lower limb or spine
* Developmental disorder in the patients history

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Length of the femoral mechanical axis (femur length) - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters, including:
  • Length of the tibial mechanical axis (tibia length) - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • The length of the lower limb (limb length) - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femoral head diameter - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Neck length (the distance between the centre of the femoral head and the proximal diaphyseal axis, when following the axis of the femoral neck) - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Neck shaft angle, aka the collodiaphyseal angle (CD angle, the angle between the femoral neck axis and the proximal diaphysis axis) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femoral offset (the distance between the centre of the femoral head and the closest point of the femoral shaft axis) - mm
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Mechanical tibiofemoral angle (mTFA, the angle between the mechanical axis of the femur (which passes from the femoral head through the centre of the distal femur) and the mechanical axis of the tibia (from the centre of the proximal tibia to the middle of the ankle) in the frontal plane of knee (convention dictates that in the varus position angles are negative, and in valgus positive) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Sagittal tibiofemoral angle (sTFA, the angle between the femural and tibial mechanical axis in the sagittal plane) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femoral mechanical axis-femoral shaft angle (FM-FS, the angle between the mechanical and anatomical axis of the femur in the frontal plane of the knee) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femur mechanical angle (FMA, the angle between the femoral mechanical axis and the tangent of the femoral condyles medially) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Tibial mechanical angle (TMA, the angle between tibial mechanical axis and the tangent of the tibia plateau medially) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femoral torsion (the angle between the femoral neck axis and the posterior condylar line projected on a plane perpendicular to the mechanical axis of the femur) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Tibial torsion (the angle between the transmalleolar and transcondylar axis projected on a plane perpendicular to the mechanical axis of the tibia) - degrees
3D reconstruction with 15 anatomical and biomechanical parameter of the lower limb | 6 months
  Based on the stereo radiographs, SterEOS 3D reconstruction will be done. The SterEOS software calculates automatically 15 parameters including:
  • Femorotibial rotation (the angle between the posterior condylar line of the femur and tibia) - degrees

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Schlegl, M.D., Ph.D., Principal Investigator — University of Pecs Medical School, Department of Orthopaedics
Locations (1):
- Ádám Schlégl, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
If the approval of the participants make it possible, the whole dataset will be published.